CLINICAL TRIAL: NCT01891721
Title: Evaluating Two Types of Cognitive Training in Veterans With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-015-12F
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: cognitive training; schizophrenia; mismatch negativity; cognition; functional capacity; EEG
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Specific Perceptual Training - Brain Fitness Program (BFP) (Experimental): In each session, participants will work on 4 of the 6 BFP exercises (15 min per exercise). Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Interventions: Behavioral: Brain Fitness Program (BFP)
- Broad Cognitive Training - Cognitive Package (Cogpack) (Experimental): In each session, participants will work on a different subset of 4 to 6 Cogpack exercises. Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Interventions: Behavioral: Cognitive Package (Cogpack)
- Control Treatment - Commercial Computer Games (Sporcle) (Active Comparator): In each session, participants will play between 8 and 16 games (1 to 15 min per game). Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Interventions: Behavioral: Commercial Computer Games (Sporcle)

INTERVENTIONS:
Behavioral: Brain Fitness Program (BFP) — This computerized "bottom-up" cognitive intervention is designed to improve the speed and accuracy of auditory information processing through increasingly more difficult stimulus recognition, discrimination, sequencing, and memory tasks under conditions of close attentional control, high reward, and novelty. BFP consists of 6 exercises. Stimuli across the exercises are chosen such that they span the acoustic and organizational structure of speech, from very simple acoustic stimuli and tasks to complex manipulations of continuous speech. The exercises adaptively progress based on the subject's individual performance during a training session and become more challenging as the subject's abilities improve. Participants will work with 4 of the 6 exercises (15 min per exercise) in each session.
  Arms: Specific Perceptual Training - Brain Fitness Program (BFP)
Behavioral: Cognitive Package (Cogpack) — This computerized "top-down" cognitive intervention is designed to provide training across a broad range of cognitive functions. Cogpack consists of domain-specific exercises aimed at training specific cognitive areas (attention, working memory, verbal and visual memory, executive functioning, reasoning, language) and non-domain-specific exercises that require the use of several functions at a time. Cogpack includes low-level cognitive exercises (i.e., scanning, hand-eye coordination, and psychomotor speed) that will not be included in this protocol to better separate bottom-up from top-down training interventions. There will be a total of 34 exercises and variants of the same exercises with different levels of difficulty. In each session, participants will work on a different subset of 4 to 6 exercises.
  Arms: Broad Cognitive Training - Cognitive Package (Cogpack)
Behavioral: Commercial Computer Games (Sporcle) — Sporcle computer games will be used as a "placebo" treatment to control for the effects of computer exposure, contact with research personnel, time spent being cognitively active, and financial compensation for participation. The games cover trivia-type questions about geography, entertainment, science, history, literature, sports, movies, etc. Subjects will receive the same amount of attention from staff members and the same monetary reinforcements as participants in the experimental treatment groups. They will also complete 3 hours of "training" per week over 12 weeks, for a total of 36 hours.
  Arms: Control Treatment - Commercial Computer Games (Sporcle)

SUMMARY:
Cognitive dysfunction is a major contributor to the poor community outcome of individuals with schizophrenia. Developing more effective cognitive remediation interventions is imperative to improve the daily lives of affected subjects and reduce the disability of this illness. The goal of this clinical trial is to evaluate two types of cognitive training approaches to determine which one is more beneficial for individuals with schizophrenia. This study also uses electrophysiological techniques to gain a better understanding of the mechanisms involved in cognitive remediation. Findings from this study will provide information about how to design the most optimally efficient cognitive training intervention to improve the cognitive and social functioning of patients with severe mental illness.

DETAILED DESCRIPTION:
Schizophrenia is a disorder that affects both higher-level neurocognitive operations (e.g., verbal memory, executive functioning) and lower-level perceptual processes (e.g., auditory processing). These deficits contribute to the poor community outcome and severe functional disability seen in patients. Effectively treating the cognitive dysfunction associated with this illness is important to achieve improvements in daily functioning. Recent meta-analytic studies report that cognitive training in schizophrenia has a moderate effect-size impact on cognitive functioning and a lower impact on daily functioning. However, most training interventions for schizophrenia have only targeted higher-order cognitive processes. A few recent interventions have targeted basic perceptual processing and shown that auditory and visual perceptual abilities can be trained and improved in patients with schizophrenia. These findings suggest that basic perceptual processing may be an ideal target for intervention. At this point, it is still unclear whether a neuroplasticity-based, bottom-up intervention is more effective than an intervention that targets top-down functions like attention, working memory, and executive functioning.

This clinical trial will contrast a bottom-up intervention targeting basic auditory processes and a top-down intervention targeting higher-order cognitive functions, compared with a control condition, in Veterans with schizophrenia. These interventions will be assessed by their effects on representative measures from three outcome domains: 1) neurocognition, 2) electroencephalography (EEG), and 3) functional capacity. Participants will be randomly assigned to the bottom-up auditory training, top-down cognitive training, or control treatment (commercial computer games). All treatments will be administered three times a week (1 hour each) for 12 weeks. A comprehensive battery of cognitive, electrophysiological, and functional measures will be administered at baseline, 6 weeks, and at completion of treatment. The investigators will enroll 120 Veterans with schizophrenia or schizoaffective disorder across the 5 years of the study.

This study will determine which training approach leads to the largest magnitude of improvement in neurocognition, functional capacity, and neural functioning measured with EEG. Moreover, it will shed light on the neural mechanisms underlying the response to training. By determining whether it is more beneficial to treat lower-level perceptual processes or higher-level cognitive functions, the results of this project will inform future recovery-based cognitive remediation interventions for Veterans with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder
* Between 25 and 65 years of age
* Estimated premorbid inteIligence quotient (IQ) > 70 (based on reading ability)
* Understand spoken English sufficiently to comprehend the consent form
* Clinically stable (i.e., no inpatient hospitalization in the 3 months, no changes in psychiatric medications in the 6 weeks, and no changes in housing in the 2 months, prior to enrollment)

Exclusion Criteria:

* Documented history of mental retardation or severe learning disability
* Clinically significant neurological disease as determined by medical history (e.g., epilepsy, stroke)
* History of serious head injury with loss of consciousness greater than 1 hour and concomitant neuropsychological sequelae
* Meeting DSM-IV criteria for drug or alcohol dependence during the 6 months, or abuse during the month preceding study enrollment

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Jahchan, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (2):
- United States (2):
  - Local Board and Care Facilities, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adcock RA, Dale C, Fisher M, Aldebot S, Genevsky A, Simpson GV, Nagarajan S, Vinogradov S. When top-down meets bottom-up: auditory training enhances verbal memory in schizophrenia. Schizophr Bull. 2009 Nov;35(6):1132-41. doi: 10.1093/schbul/sbp068. Epub 2009 Sep 10. PMID 19745022
- [Background] Medalia A, Choi J. Cognitive remediation in schizophrenia. Neuropsychol Rev. 2009 Sep;19(3):353-64. doi: 10.1007/s11065-009-9097-y. Epub 2009 May 15. PMID 19444614
- [Background] Popov T, Jordanov T, Rockstroh B, Elbert T, Merzenich MM, Miller GA. Specific cognitive training normalizes auditory sensory gating in schizophrenia: a randomized trial. Biol Psychiatry. 2011 Mar 1;69(5):465-71. doi: 10.1016/j.biopsych.2010.09.028. Epub 2010 Nov 18. PMID 21092939
- [Background] Green MF, Kern RS, Braff DL, Mintz J. Neurocognitive deficits and functional outcome in schizophrenia: are we measuring the "right stuff"? Schizophr Bull. 2000;26(1):119-36. doi: 10.1093/oxfordjournals.schbul.a033430. PMID 10755673
- [Background] Fisher M, Holland C, Merzenich MM, Vinogradov S. Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia. Am J Psychiatry. 2009 Jul;166(7):805-11. doi: 10.1176/appi.ajp.2009.08050757. Epub 2009 May 15. PMID 19448187
- [Background] Light GA, Braff DL. Mismatch negativity deficits are associated with poor functioning in schizophrenia patients. Arch Gen Psychiatry. 2005 Feb;62(2):127-36. doi: 10.1001/archpsyc.62.2.127. PMID 15699289

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants were excluded from the study before being randomized to groups: 4 for not meeting inclusion criteria and 2 for not wanting to participate.
Groups:
- Specific Perceptual Training - Brain Fitness Program (BFP): In each session, participants worked on 4 of the 6 BFP exercises (15 min per exercise). Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Brain Fitness Program (BFP): This computerized "bottom-up" cognitive intervention is designed to improve the speed and accuracy of auditory information processing through increasingly more difficult stimulus recognition, discrimination, sequencing, and memory tasks under conditions of close attentional control, high reward, and novelty. BFP consists of 6 exercises. Stimuli across the exercises are chosen such that they span the acoustic and organizational structure of speech, from very simple acoustic stimuli and tasks to complex manipulations of continuous speech. The exercises adaptively progress based on the subject's individual performance during a training session and become more challenging as the subject's abilities improve.
- Broad Cognitive Training - Cognitive Package (Cogpack): In each session, participants worked on a different subset of 4 to 6 Cogpack exercises. Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Cognitive Package (Cogpack): This computerized "top-down" cognitive intervention is designed to provide training across a broad range of cognitive functions. Cogpack consists of domain-specific exercises aimed at training specific cognitive areas (attention, working memory, verbal and visual memory, executive functioning, reasoning, language) and non-domain-specific exercises that require the use of several functions at a time. Cogpack includes low-level cognitive exercises (i.e., scanning, hand-eye coordination, psychomotor speed) that will not be included in this protocol to better separate bottom-up from top-down training interventions. There will be a total of 34 exercises and variants of the same exercises with different levels of difficulty.
- Control Treatment - Commercial Computer Games (Sporcle): In each session, participants played between 8 and 16 games (1 to 15 min per game). Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Commercial Computer Games (Sporcle): Sporcle computer games were used as a "placebo" treatment to control for the effects of computer exposure, contact with research personnel, time spent being cognitively active, and financial compensation for participation. The games cover trivia-type questions about geography, entertainment, science, history, literature, sports, movies, etc. Subjects received the same amount of attention from staff members and the same monetary reinforcements as participants in the experimental treatment groups. They also completed 3 hours of "training" per week over 12 weeks, for a total of 36 hours.
Period: Overall Study
Arm/Group | Specific Perceptual Training - Brain Fitness Program (BFP) | Broad Cognitive Training - Cognitive Package (Cogpack) | Control Treatment - Commercial Computer Games (Sporcle)
Started | 39 | 40 | 20
Completed | 29 | 35 | 19
Not Completed | 10 | 5 | 1
Not completed — Lost to Follow-up | 10 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Broad Cognitive Training - Cognitive Package (Cogpack): In each session, participants worked on a different subset of 4 to 6 Cogpack exercises. Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Cognitive Package (Cogpack): This computerized "top-down" cognitive intervention is designed to provide training across a broad range of cognitive functions. Cogpack consists of domain-specific exercises aimed at training specific cognitive areas (attention, working memory, verbal and visual memory, executive functioning, reasoning, language) and non-domain-specific exercises that require the use of several functions at a time. Cogpack includes low-level cognitive exercises (i.e., scanning, hand-eye coordination, psychomotor speed) that were not included in this protocol to better separate bottom-up from top-down training interventions. There was a total of 34 exercises and variants of the same exercises with different levels of difficulty.
- Total: Total of all reporting groups
Arm/Group | Specific Perceptual Training - Brain Fitness Program (BFP) | Broad Cognitive Training - Cognitive Package (Cogpack) | Control Treatment - Commercial Computer Games (Sporcle) | Total
Number analyzed (Participants) | 39 | 40 | 20 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.59 (9.44) | 51.05 (9.42) | 51.0 (9.54) | 51.18 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 6 | 22
  Male | 32 | 31 | 14 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 4 | 14
  Not Hispanic or Latino | 33 | 35 | 16 | 84
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 14 | 11 | 46
  White | 13 | 23 | 9 | 45
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 40 | 20 | 99
MCCB neurocognition composite [Mean (Standard Deviation); unit: units on a scale] — The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) was used to assess basic cognition. It includes tests representing 6 separable cognitive domains. The MCCB composite score (average of 6 domain t-scores) served as the primary cognitive outcome measure. Minimum and maximum values are 20 and 68. Higher scores mean a better outcome.
  units on a scale | 42.52 (8.75) | 41.57 (8.41) | 41.18 (8.70) | 41.76 (8.62)
UPSA total [Mean (Standard Deviation); unit: units on a scale] — The University of California San Diego (UCSD) Performance-based Skills Assessment (UPSA) was used to assess functional capacity. The UPSA total score served as a secondary functional outcome measure. Minimum and maximum values are 40 and 100. Higher scores mean a better outcome.
  units on a scale | 74.85 (10.73) | 74.27 (11.72) | 77.25 (13.99) | 75.46 (12.15)
MMN amplitude [Mean (Standard Deviation); unit: units on a scale] — A Mismatch Negativity (MMN) Paradigm was used to assess basic auditory processing. MMN amplitude was measured as the mean voltage in the 145-200 ms latency range at pooled frontocentral electodes. Minimum and maximum values are -8 and +2 microvolts. More negative scores mean a better outcome.
  units on a scale | -2.21 (2.12) | -2.25 (1.69) | -2.18 (2.18) | -2.21 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Neurocognition
Description: The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) was used to assess basic cognition. It includes tests representing 6 separable cognitive domains. The MCCB composite score (average of 6 domain t-scores) served as the primary cognitive outcome measure. Minimum and maximum values are 20 and 68. Higher scores mean a better outcome.
Time Frame: Within one week of training completion
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Specific Auditory Training - Brain Fitness Program (BFP): In each session, participants worked on 4 of the 6 BFP exercises (15 min per exercise). Duration of training is 1 hour per day, 3 days per week, for 12 weeks, for a total of 36 hours.
  Brain Fitness Program (BFP): This computerized "bottom-up" cognitive intervention is designed to improve the speed and accuracy of auditory information processing through increasingly more difficult stimulus recognition, discrimination, sequencing, and memory tasks under conditions of close attentional control, high reward, and novelty. BFP consists of 6 exercises. Stimuli across the exercises are chosen such that they span the acoustic and organizational structure of speech, from very simple acoustic stimuli and tasks to complex manipulations of continuous speech. The exercises adaptively progress based on the subject's individual performance during a training session and become more challenging as the subject's abilities improve.
Arm/Group | Specific Auditory Training - Brain Fitness Program (BFP) | Broad Cognitive Training - Cognitive Package (Cogpack) | Control Treatment - Commercial Computer Games (Sporcle)
Number analyzed (Participants) | 29 | 35 | 19
score on a scale | 42.02 (7.96) | 41.92 (8.47) | 41.94 (8.72)

2. Secondary Outcome: Electroencephalography (EEG)
Description: A Mismatch Negativity (MMN) Paradigm was used to assess basic auditory processing. MMN amplitude was measured as the mean voltage in the 145-200 ms latency range at pooled frontocentral electodes. Minimum and maximum values are -8 and +2 microvolts. More negative scores mean a better outcome.
Time Frame: After 6 weeks of training and within one week of training completion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Specific Auditory Training - Brain Fitness Program (BFP) | Broad Cognitive Training - Cognitive Package (Cogpack) | Control Treatment - Commercial Computer Games (Sporcle)
Number analyzed (Participants) | 29 | 35 | 19
units on a scale
  MMN at 12 weeks | -2.04 (1.77) | -2.17 (1.86) | -2.09 (1.87)
  MMN at 6 weeks | -1.78 (1.76) | -2.16 (1.83) | -2.21 (1.90)

3. Secondary Outcome: Functional Capacity
Description: The University of California San Diego (UCSD) Performance-based Skills Assessment (UPSA) was used to assess functional capacity. The UPSA total score served as a secondary functional outcome measure. Minimum and maximum values are 40 and 100. Higher scores mean a better outcome.
Time Frame: Within one week of training completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Specific Auditory Training - Brain Fitness Program (BFP) | Broad Cognitive Training - Cognitive Package (Cogpack) | Control Treatment - Commercial Computer Games (Sporcle)
Number analyzed (Participants) | 29 | 35 | 19
score on a scale | 76.50 (10.59) | 75.96 (11.25) | 76.77 (11.51)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Specific Perceptual Training - Brain Fitness Program (BFP) | Broad Cognitive Training - Cognitive Package (Cogpack) | Control Treatment - Commercial Computer Games (Sporcle)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 2/39 | 2/40 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Specific Perceptual Training - Brain Fitness Program (BFP) (N=39) | Broad Cognitive Training - Cognitive Package (Cogpack) (N=40) | Control Treatment - Commercial Computer Games (Sporcle) (N=20)
Other (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) — Patient reported exacerbation of psychotic symptoms likely due to underlying diagnosis not to study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT01891721/Prot_SAP_000.pdf